CLINICAL TRIAL: NCT03324828
Title: Double-blind Randomized Clinical Trial to Compare Presurgery Anxiolysis in Children Treated With Hydroxyzine Versus Non-pharmacological Intervention (Distractoria Technique Clown)
Brief Title: Presurgery Anxiolysis in Children Treated With Hydroxyzine Versus Non-pharmacological Intervention (Distractoria Technique Clown)
Acronym: SONRISA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Esther Aleo Lujan, Esther Aleo Lujan, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SONRISA
Record Dates: First submitted 2017-10-21; First posted 2017-10-30 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Anxiety
Keywords: anxiety; surgery; clown
MeSH Terms: conditions — Anxiety Disorders | interventions — Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clowns: outcomes assesor Hidroxicine: participant, care provider, investigator and outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hydroxyzine+no clowns (Active Comparator): Patients will receive hydroxyzine solution and no additional intervention
  Interventions: Drug: Hydroxyzine
- Hydroxyzine+clowns (Experimental): Patients will receive hydroxyzine solution and clowns intervention
  Interventions: Drug: Hydroxyzine; Other: Clowns intervention
- Placebo+clowns (Active Comparator): Patients will receive placebo solution and clowns intervention
  Interventions: Other: Clowns intervention
- Placebo+no clowns (No Intervention): Patients will receive placebo solution and no additional intervention

INTERVENTIONS:
Drug: Hydroxyzine — Hydroxyzine solution
  Arms: Hydroxyzine+clowns; Hydroxyzine+no clowns
Other: Clowns intervention — Clowns intervention
  Arms: Hydroxyzine+clowns; Placebo+clowns

SUMMARY:
This study evaluate the change in preoperative anxiety, baseline (M1) and pre-induction anxiety levels (M3), as shown by children undergoing MAS determined by the m-YPAS scale in the different APO management groups.Patients will be allocated in one of this four groups: hydroxyzine+clown; hydroxyzine alone, clowns alone or nothing

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 16 years old
* Patients with programmed major ambulatory surgery.
* Assessment of anesthetic risk ASA I-II.
* Informed consent signed by their legal authorized representatives.
* No antihistaminic allergies.
* Assent signed by children between 12 and 16 years old.

Exclusion Criteria:

* Patients with previous surgeries.
* Anesthetic risk ASA more than II.
* Patients with hypersensitivity to the active substance, to any of the excipients, to cetirizine, to other piperazine derivatives, to aminophylline or etilenamida
* Patients with porphyria
* Patients with known QT prolongation, either congenital or acquired
* Patients with known risk factors for QT prolongation including a pre-existing cardiovascular disease, previous electrolyte imbalances, family history of sudden cardiac death, significant bradycardia and concomitant use of drugs with potential known to produce QT prolongation and / or induce Torsades de Pointes.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
m-YPAS | Anxiety in the operation room (average 60 minutes from the begining of the study)
  Yale Preoperative Anxiety Scale (mYPAS)

SECONDARY OUTCOMES:
m-YPAS | Anxiety when the patient arrives at operation room (average 45 minutes from the begining of the study)
  Yale Preoperative Anxiety Scale (mYPAS)
Cortisol level (blood) | Just before starting surgery (average 75 minutes from the begining of the study)
  cortisol blood test
Cortisol level (salive) | when the patient arrives at operation room(average 45 minutes from the begining of the study)
  cortisol blood test
Anesthesia induction | Just before starting surgery (average 75 minutes from the begining of the study)
  Anesthesia induction according to the checklist

CONTACTS AND LOCATIONS:
Overall Officials: Esther Aleo Lujan, MD, Study Chair — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

REFERENCES:
- [Derived] Aleo E, Picado AL, Abancens BJ, Soto Beauregard C, Tur Salamanca N, Esteban Polonios C, Torrejon MJ, Perrino CG, Rivas A, Arias E, Rodriguez D, Rivas MA, Rojo MLR, Garcia PF, Alarcon JR, San Pedro de Urquiza B. Evaluation of the Effect of Hydroxyzine on Preoperative Anxiety and Anesthetic Adequacy in Children: Double Blind Randomized Clinical Trial. Biomed Res Int. 2021 Nov 11;2021:7394042. doi: 10.1155/2021/7394042. eCollection 2021. PMID 34805403
- [Derived] Aleo Lujan E, Lopez-Picado A, Rivas A, Joyanes Abancens B, Rodriguez Rojo ML, Fernandez Garcia P, Soto Beauregard C, Rodriguez Alarcon J, Gonzalez Perrino C, San Pedro de Urquiza B, Arias E, Rodriguez D, Esteban Polonio C, Torrejon MJ. Pre-operative anxiolysis in children through a combined pharmacological therapy with hydroxyzine and a non-pharmacological distraction technique with a clown (SONRISA): study protocol for randomised double-blind clinical trial. Trials. 2020 Jan 2;21(1):1. doi: 10.1186/s13063-019-3906-2. PMID 31898511